CLINICAL TRIAL: NCT04701255
Title: Difference in Postoperative Total Wavefront Pattern Between Aspheric and Negative Spherical Aberration Intraocular Lenses Implanted in Cataract Surgery
Brief Title: Postoperative Total Wavefront Pattern Between Two Types of Intraocular Lenses Implanted in Cataract Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aya Ghonaim, resident of ophthalmology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 336-2020
Record Dates: First submitted 2021-01-06; First posted 2021-01-08 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Cataract
Keywords: aberration-free; negative spherical aberration; phacoemulsification; intraocular lens; wavefront
MeSH Terms: conditions — Cataract | interventions — Phacoemulsification; Lens Implantation, Intraocular

STUDY DESIGN:
Intervention Model Description: 40 human eyes undergoing phacoemulsification with intraocular lens implantation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- aberration-free IOL (Experimental): 20 human eyes with aberration-free intraocular lens Implantation after phacoemulsification cataract surgery
  Interventions: Procedure: phacoemulsification with intraocular lens implantation; Device: ocular aberrometer assesment
- negative spherical aberration IOL (Active Comparator): 20 human eyes with negative spherical aberration intraocular lens Implantation after phacoemulsification cataract surgery
  Interventions: Procedure: phacoemulsification with intraocular lens implantation; Device: ocular aberrometer assesment

INTERVENTIONS:
Procedure: phacoemulsification with intraocular lens implantation — treatment of cataract by phacoemulsification procedure and implantation of different types of IOLs.
Device: ocular aberrometer assesment — evaluate total ocular wavefront, corneal wavefront & internal wavefront (High order aberrations ) post operative by corneal tomography and aberrometer

SUMMARY:
With the advancement of cataract eye surgery and wavefront sensors, the previously unquantifiable refractive measurements have been identified and the high order aberrations have shown their effect on high resolution imaging.

In the human phakic eye, the shape of the normal cornea induces average positive spherical aberration and remains unchanged over time, whereas the crystalline lens has a negative spherical aberration. As a result, overall spherical aberration in the young eye is low.

However, the compensation slowly decreases with the aging lens and is fully lost after cataract extraction and implantation of a standard intraocular lens.

Optical studies showed that conventional biconvex spherical intraocular lenses add their intrinsic positive spherical aberration to the positive spherical aberration of the cornea resulting in image imperfection and blur. As a useful side effect, this also increases the depth of focus -often referred to as pseudo-accommodation.

New Aspheric intraocular lenses designs currently in use impart negative spherical aberration, about 0.17 to 0.20 microns of negative spherical aberration. This added negative spherical aberration partially corrects the average amount of corneal positive spherical aberration & compensate for its effect. Our study will include (FocusForce foldable aspheric intraocular lens, Bausch & Lomb, New Jersey, USA) as an example of this type of negative spherical aberration intraocular lenses.

In order to improve retinal image quality without compromising depth of field, or introducing other aberrations, aberration-free aspheric intraocular lenses were developed with no inherent spherical aberration.

The other intraocular lens targeted in our study (Akreos AO Microincision lens, Bausch & Lomb, New Jersey, USA) is an example of this type of IOLs.

DETAILED DESCRIPTION:
A customized correction for the individual eye seems to be the most promising solution for tailored correction of spherical aberration.

On the other hand, Wave front analysis of the ocular optical system has increased our knowledge of the aberrations in the eye. The importance of measuring optical aberrations lies not only in the presence of natural aberrations in the human eye, but also in its usefulness for evaluating individual surgical outcomes. By using Zernike polynomials, the aberrations of the ocular system can be characterized. Zernike coefficients of the higher-order aberrations can be derived from corneal topographic data. And for those generated by the whole optical system of the eye can be derived from aberrometry.

With current small-incision cataract surgery, it has been reported that the average postoperative corneal topography does not differ significantly from average preoperative corneal topography, so in our study we will focus on the ocular & internal wave front changes.

With the high resolution pyramid wavefront sensor incorporated in (SCHWIND PERAMIS®, topography and Aberrometry, Kleinostheim, Germany) we will evaluate and compare the total ocular wave front and the corneal wave front in our study to identify and estimate the internal aberrations . This new sensor uses an extended source instead of a point-like source avoiding in this manner the oscillation of the pyramid.

SCHWIND PERAMIS evaluates the ocular wave front aberrations with 45,000 measuring points - without any overlap and with clear assignment of each point & records 33 images per second and automatically selects the image with the best measurement. Together with real-time measurement, this ensures a new level of detail resolution and precision. SCHWIND PERAMIS can also be used to compare a patient's corneal and ocular wave front data. The direct comparison provides information about whether a visual defect is located on the surface of the cornea or within the eye itself, thus allowing us to identify and evaluate internal aberrations.

ELIGIBILITY:
Inclusion Criteria:

1-All patients with written informed consent, between the age of 21 -75 years who will undergo phacoemulsification procedure with intraocular lens implantation of one of the targeted lenses in the study

Exclusion Criteria:

1. Previous corneal intervention or refractive surgery.
2. Persistent Corneal edema (epithelial or stromal).
3. Co-existing corneal pathology.
4. Ocular surface disease & Dry eye syndrome.
5. Posterior capsular opacity .
6. Anterior capsular contraction (phimosis).
7. Ocular inflammation.
8. Co-existing Vitreoretinal diseases.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-11-09 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Corneal, Ocular, and Internal spherical aberrations | 1 month postoperative
  assessment of ocular, corneal & internal wavefront by aberrometer & corneal tomography

SECONDARY OUTCOMES:
corneal wavefront changes | 1 month postoperative
  • Compare pre-operative and post-operative corneal spherical aberrations of every patient and evaluate any significant changes.
near vision addition | 1 month postoperative
  the plus lenses needed to be add to correct near vision which reflect the depth of focus of the IOL implanted

CONTACTS AND LOCATIONS:
Overall Officials: Aya G Ibrahim, MBBCh, Principal Investigator — Dar El Oyoun ophthalmology hospital
Locations (1):
- facultyof medicine, Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No